CLINICAL TRIAL: NCT04139200
Title: The Long-term Effects of a Tele Coaching Intervention in Patients With COPD: a Randomized Controlled Trial
Brief Title: Long-term Activity Coaching in Patients With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: University Ghent (Other)
Responsible Party: Principal Investigator, Thierry Troosters, Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S62902
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: COPD
Keywords: Physical activity; Tele coaching
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Participant
Masking Description: Patients in the control group will receive a sham version of the smartphone application. Patients are unaware of the difference between the coaching programs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Type 1 tele coaching group (Experimental): Coaching with daily interaction with the coaching application, based on a adaptive physical activity goal
  Interventions: Behavioral: Type 1 physical activity tele coaching intervention
- Type 2 tele coaching group (Sham Comparator): Coaching with fixed physical activity goal and limited interaction with the smartphone application
  Interventions: Behavioral: Type 2 physical activity tele coaching intervention

INTERVENTIONS:
Behavioral: Type 1 physical activity tele coaching intervention — A) Education about the importance of PA. During a one-to-one interview with the coach motivation, self-efficacy, barriers, favorite activities and strategies to become more active are discussed. B) Step counter providing direct feedback. C) A smartphone with a project-tailored application. The application provides automated coaching by displaying an activity goal (number of steps) and feedback on a daily basis. The feedback comes with a graphical presentation. Patients' targets are automatically revised weekly. The aim is to progressively increase the PA during the 12 weeks period and maintain afterwards. D) Telephone contacts triggered in the case of non-compliance with wearing the step counter, failure to transmit data, failure to progress or change in medication. Coaches are alerted by a note at the coaches' backend to take contact with the patient if needed.
  Arms: Type 1 tele coaching group
Behavioral: Type 2 physical activity tele coaching intervention — A) Education about the importance of PA. During a one-to-one interview with the investigator, patients will receive a personal goal (expressed in steps/day), based on their individual exercise capacity. B) A step counter providing direct feedback. C) A smartphone with a project-tailored application. The application receives the step data of the patient and asks on a weekly basis about the patient's change in medication. The application does provide a graph showing the steps the patient took and presents a general activity plan including their personal goal (which stays the same throughout the entire intervention period). D) Telephone contacts triggered in the case of change in medication. Coaches are alerted by a note at the coaches' backend to take contact with the patient if needed.
  Arms: Type 2 tele coaching group

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a leading cause of mortality and morbidity around the world. Studies revealed that patients with COPD are less active than age-matched healthy controls and activity level decreases with disease severity. Higher levels of physical activity is related to important health-related outcomes, such as lower mortality rate and hospital admissions. Additionally, increasing physical activity is related with substantial health benefits. Patients with COPD have a higher risk of developing insulin resistance, hypertension, dyslipidemia, osteopenia, leading to chronic diseases such as coronary heart disease, type 2 diabetes and osteoporosis, which have been related to physical inactivity in the healthy population. Moreover, physical inactivity has been related to the occurrence of comorbidities in patients with COPD. Therefore, improving physical activity levels is a recommended treatment in the disease management in all patients with COPD and is implemented in the recent GOLD guidelines for all patients with COPD, regardless of the disease severity.

The research group investigated the effect of a 3-month semi-automatic tele-coaching intervention on physical activity levels in patients with COPD. The tele coaching intervention led to a significant improvement on physical activity in the intervention group. Although this trial showed positive results on physical activity, further research is needed, mainly to investigate the long-term (12 months) effectiveness of such interventions and the added value of a smartphone application on top of a simple step counter providing feedback. Additionally, since physical activity is related to the development of comorbidities, the investigators aim to explore the influence of improving physical activity levels on the occurrence of cardiovascular, metabolic and musculoskeletal comorbidities. Finally, this study will explore baseline characteristics (such as social support, self-efficacy, dynamic hyperinflation, etc.) that can predict success in this intervention.

DETAILED DESCRIPTION:
The aims of the present study are:

1. primary objective: To investigate the changes in physical activity after a 12-month tele coaching intervention (including individualized goal setting, feedback, motivational contacts with coach and a step counter providing direct feedback), compared to a sham group receiving a light coaching intervention (feedback from step counter and static goal setting, without additional motivation or contact with the coach).
2. secondary objectives:

A. Investigate the effect of a 12-month tele coaching intervention on exercise capacity, muscle force, quality of life, physical activity from a patient's perspective, dyspnea-related fear and comorbidities.

B. Confirming previous findings on short-term effects (or lack of effect) of the tele coaching intervention on physical activity, exercise capacity and quality of life, assessed at 6 months.

C. Identifying possible baseline characteristics that are determinants of the change in physical activity after the 12-month tele coaching intervention.

D. Investigating the association between the pattern in vital signs (including physical activity, resting heart rate, heart rate variability, heart rate recovery, oxygen saturation, respiratory rate) as measured by a wearable and the onset of an exacerbation.

E. To explore the relation between dynamic hyperinflation as measured during the six-minutes walk test, physical activity measured at baseline and change in physical activity as result of the intervention.

F. Investigate the effect of an acute exacerbation on functional performance (only in Ghent).

G. Investigate the association between a change in physical activity and autonomic function (only in Ghent).

H. Validity and reliability of wearable devices to measure autonomic function, respiratory rate and oxygen saturation (only in Ghent).

Therefore, the study will include stable patients with COPD (post bronchodilator FEV1/FVC < 0.70) with no moderate or severe exacerbations in the past month, across all disease severities.

For patients in UZ Leuven and UZ Ghent, the study will consists of 4 clinical visits:

* Visit 1 screening visit
* Visit 2: randomization visit, scheduled 1-2 weeks after visit 1
* Visit 3: short term follow-up visit, scheduled 6 months after visit 2
* Visit 4: long-term follow-up visit, scheduled 12 months after visit 2

Only for patients in UZ Ghent: to investigate the effect of an acute COPD exacerbation on functional performance, an additional visit will take place when the patient experiences an exacerbation after the first 6 months of the study. This visit will take place as soon as possible and maximally 14 days after onset of the symptoms.

If the patient does not experience an exacerbation during the first year of the study, the patient will be followed-up until occurrence of the first exacerbation or up to 30 months (whichever occurs first) with intermediate visits at 18 months and 24 months.

All patients included in the study will be randomized in either the intervention group or sham group:

* A multicomponent tele coaching intervention that consists of 1) education about the importance of physical activity and a one-to-one interview with the coach discussing the motivation and barriers to be active, 2) a step counter providing direct feedback, 3) application installed on a smartphone providing an adaptive goal and daily and weekly feedback and 4) contact with the coach if the patient is not compliant with the intervention, not increasing physical activity or when the patient reports a change in medication. The patient is asked to have a daily interaction with the smartphone application.
* A sham intervention that consist of 1) education about the importance of physical activity and a personal (fixed) goal expressed in terms of steps. The patient is asked to try to reach this goal, 2) a step counter providing direct feedback, 3) application installed on a smartphone only displaying a graph with the activity of the present week and the personal (fixed) goal, 4) contact with the coach if the patient reports a change in medication. The patient is asked to have at least a weekly interaction with the application.
* Only in UZ Ghent: in case of extended follow-up after 12 months, patients will receive the multicompenent tele coaching intervention after 12 months of inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with COPD (GOLD criteria post bronchodilator FEV1/FVC < 0.70)
2. Patients under medical follow-up of a respiratory physician or general practitioner with no moderate (ambulatory treated) and/or severe (requiring a hospital admission) exacerbation in the past month
3. Older than 40 years old
4. Smoking history with more than 10 pack years

Exclusion Criteria:

1. The presence of orthopedic or other problems not allowing an increase in physical activity levels
2. Unable to learn to work with a new electronic device (e.g. smartphone), as judged by the investigator
3. Underwent lung transplantation or active on the lung transplantation list
4. Involved in or planned to start with a structured multidisciplinary rehabilitation program

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Daily number of steps at 12 months | 12 months
  Change in daily mean step count 12 months post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.

SECONDARY OUTCOMES:
Daily number of steps at 6 months | 6 months
  Change in daily mean step count 6 months post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Minutes per day spent in at least moderate intense activities | 6 months and 12 months
  Change in minutes per day spent in at least moderate intense activities 6 and 12 months post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Mean walking time per day | 6 months and 12 months
  Change in mean daily walking time 6 and 12 months post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Mean sedentary time per day | 6 months and 12 months
  Change in mean sedentary time 6 and 12 months post randomization in the intervention group as compared to the control group. Physical activity will be objectively measured for 1 week using a tri-axial accelerometer validated for use in patients with COPD. At least 4 valid weekdays (> 8 hours of wearing time during waking hours) is necessary to label the physical activity measurement as valid.
Exercise capacity | 6 months and 12 months
  Change in six-minutes walk distance 6 and 12 months post randomization in the intervention group as compared to the control group. The six-minutes walk test will be performed with standardized encouragement to assess patients' functional exercise capacity. The best of two measurements will be used.
Quadriceps force | 6 months and 12 months
  Change in quadriceps force 6 and 12 months post randomization in the intervention group as compared to the control group. The quadriceps isometric strength will be evaluated by a maximal voluntary contraction using the Biodex, a computerized dynamometer. Patients will be seated with a 90° hip and 60° knee flexion. The best of 4 measurements will be taken into analysis as the maximal force capacity of the lower limb.
Health status | 6 and 12 months
  Change in health status 6 and 12 months post randomization in the intervention group as compared to the control group. Health status will be measured by COPD assessment test (CAT), a validated, 8-item questionnaire to assess the impact of the disease on a patient's health status. Scores range from 0 to 40, with a higher score indicating a worse health status. The minimal clinical important difference (MCID) is a change of 3 points.
Health related quality of life: CRDQ-SAS | 6 months and 12 months
  Change in health related quality of life 6 and 12 months post randomization in the intervention group as compared to the control group. Health status will be measured by Chronic Respiratory Disease Questionnaire; self-administrated standardized version (CRDQ-SAS), measuring both physical and emotional aspects of chronic respiratory disease. The questionnaire contains 20 items, spread over 4 domains (dyspnea, fatigue, emotional function and mastery). The minimal clinical important difference is reflected by a change in score of 0.5 on a 7-point scale.
Physical activity from a patients' perspective | 6 months and 12 months
  Change in physical activity from a patients' perspective 6 and 12 months post randomization in the intervention group as compared to the control group. This will be measured by PROactive tool (clinical visit version), a validated 12-item questionnaire assessing physical activity from a patient's perspective reflecting the past 7 days. The questionnaire investigates the amount of and difficulty with physical activity as perceived by the patient. The 2 domain scores (i.e. amount and difficulty) as well as the total score will be retrieved as outcomes. Subscores and total score are from 0 to 100, with higher score meaning less problems with daily life activities as reported by the patient.
Dyspnea-related fear | 6 months and 12 months
  Change in dyspnea-related fear 6 and 12 months post randomization in the intervention group as compared to the control group. This will be measured by breathlessness beliefs questionnaire (BBQ), an 17-item questionnaire investigating the dyspnea-related anxiety in patients with respiratory diseases. Score ranges from 17 to 85. Higher values indicate worse dyspnea-related fear.
Symptoms of anxiety and depression | 12 months
  Change in symptoms of anxiety and depression 12 months post randomization in the intervention group as compared to the control group. Symptoms of anxiety and depression will be measured by the Hospital Anxiety and Depression Scale (HADs). The HADs is a generic screening measure of symptoms of anxiety and depression. The HADS is a 14 item measure comprising 7 anxiety items and 7 depression items from which separate anxiety and depression sub-scale scores are calculated, ranging from 0 to 21 for both sub domains. A score of 8 or higher indicates a high possibility of anxiety / depression
Functional performance | Only in Ghent - as soon as possible and max 14 days after the occurrence of an COPD exacerbation
  To investigate the effect of an acute COPD exacerbation on functional performance, functional performance will be measured by the Short physical performance battery (SPPB), timed up and go test (TUG) and 1-minute sit-to-stand (1' STS) as soon as possible (and maximally 14 days) after onset of an exacerbation.
Autonomic function | Only in Ghent - 6 months and 12 months; additionally at 18 months and 24 months in case of extended design
  Exploring the association between change in physical activity and autonomic function. To evaluate the autonommic fuction, the patient will wear a Polar chest band with corresponding watch for 7 consecutive days (day and night). Based on this measurement we will retrieve measures on: respiratory rate; resting heart rate (heart rate during the night); heart rate variability. Data will be processed using Kubios software.
  The Polar chest band with corresponding watch will also be worn while performing the 6-minute walking test as measures of HRV during exercise and heart rate recovery (HRR). Data will be processed using Kubios software.
Autonomic symptoms | Only in Ghent - 6 months and 12 months; additionally at 18 months and 24 months in case of extended design
  Exploring the association between change in physical activity and autonomic fuction, To evaluate autonomic symptoms, autonomic symptoms will be measured by the COMPASS 31 questionnaire. This questionnaire contains six domains: orthostatic intolerance, vasomotor, secrotomotor, gastrointestinal, urinary and pupillomotor function. Total score ranges from 0 to 100, with higher score indicating more autonomic dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, Prof, Principal Investigator — KU Leuven; Heleen Demeyer, Dr, Principal Investigator — KU Leuven; Thierry Troosters, Prof, Principal Investigator — KU Leuven; Nikolaas De Maeyer, Dr, Principal Investigator — UZ Leuven; Astrid Blondeel, Principal Investigator — KU Leuven; Eric Derom, Prof.Dr., Principal Investigator — UZ Gent; Fien Hermans, Principal Investigator — U Gent
Locations (2):
- Belgium (2):
  - UZ Gent, Ghent
  - UZ Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blondeel A, Hermans F, Breuls S, Wuyts M, Everaerts S, De Maeyer N, Derom E, Janssens W, Demeyer H, Troosters T. A Long-Term Physical Activity Coaching Program for Patients with Chronic Obstructive Pulmonary Disease: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2025 Dec;211(12):2330-2339. doi: 10.1164/rccm.202501-0170OC. PMID 40700740